CLINICAL TRIAL: NCT05013164
Title: Role of Folinic Acid in Improving the Adaptive Skills and Language Impairment in Children With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Hashim Raza, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICHMultan
Record Dates: First submitted 2021-08-10; First posted 2021-08-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folinic Acid + Behavioral Therapy (Experimental): Children receiving folinic acid and behavioral therapy. Folinic Acid was given at the dose of 2mg/kg per day in two divide doses( maximum 50 mg per day) given for 12 weeks.
  Interventions: Drug: Folinic Acid
- Behavioral Therapy (No Intervention): Children received only behavioral therapy for 12 weeks.

INTERVENTIONS:
Drug: Folinic Acid — Folinic Acid was given at the dose of 2mg/kg per day in two divide doses( maximum 50 mg per day) given for 12 weeks
  Arms: Folinic Acid + Behavioral Therapy

SUMMARY:
No such study has been conducted in Pakistan so the primary objective of this study was to determine the role of folinic acid in improving the speech and adaptive skills while secondary objective was improvement of stereotype movements and hyperactivity in ASD among children aged 3 to 14 years.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders aged 3 to 14 years with diagnosis of autism spectrum disorder established by DSM-5 Criteria, Childhood Autism Rating Scale (CARS) scoring and clinical examination along with documentation of Language Impairment

Exclusion Criteria:

* All children having autism with seizure disorder, autism with serious medical illness within last 6 months or those with autism with well-defined genetic syndrome.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
To determine the role of folinic acid in improving the speech and adaptive skills among children with autism spectrum disorders | 12 weeks
  Outcome measures were based on Autism Symptoms Questionnaire (Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, et al. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Molecular Psychiatry. 2016;23(2):1-10. doi:10.1038/mp.2016.168). Primary outcome measures was language improvement and adaptive skills (gross motor development age, self-help).

SECONDARY OUTCOMES:
To dertermine improvement of stereotype movements and hyperactivity in children with autism spectrum disorders | 12 weeks
  Secondary outcome measures were improvement in stereotype movements, verbal communication, hyperactivity, peer relationship and inattention based on Autism Symptoms Questionnaire (Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, et al. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Molecular Psychiatry. 2016;23(2):1-10. doi:10.1038/mp.2016.168)

CONTACTS AND LOCATIONS:
Overall Officials: Fawwad Saleem, FCPS, Principal Investigator — ICH Multan, Pakistan
Locations (1):
- Children's Hospital and Institute of Child Health, Multan, Punjab Province, Pakistan